CLINICAL TRIAL: NCT07006051
Title: The TCU Athlete Study
Brief Title: The TCU Division I Collegiate Athlete Study
Status: Active, not recruiting | Type: Observational
Sponsor: Texas Christian University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#2023-124
Record Dates: First submitted 2025-04-08; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Orthopaedic Injuries; Concussion (Diagnosis)
Keywords: Concussion; Mild Traumatic Brain Injury; Collegiate Athlete; Orthopaedic Injury
MeSH Terms: conditions — Brain Concussion; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Collegiate Athletes: All subjects must be current NCAA Division 1 collegiate level athletes at Texas Christian University. Subject testing will include: neurocognitive tests, balance tests, jump tests, strength tests.
  Interventions: Other: Exposed group

INTERVENTIONS:
Other: Exposed group — All subjects are tested pre-season for their sport. They are then prospectively followed for orthopaedic and/or concussive injury. If injuries occur, then repeat testing is performed.
  Other Names: Exposure to Orthopaedic injury; Exposure to concussive injury

SUMMARY:
The overall objective of this study is to identify risk factors for two of the most common types of injuries in collegiate athletics - orthopedic injuries and concussion injuries.

Aim 1 of this study is to investigate risk factors for orthopedic injuries from a brief testing battery developed by the research team.

Aim 2 of this study is to investigate risk factors for concussion injuries and subsequent sequelae after returning to play from concussion from the same brief testing battery developed by the research team. Additionally, we will examine the relationships between orthopedic injuries and concussion injuries in the collegiate athlete.

Participants will participate in a pre-season battery of tests that include:

* Balance assessment
* Jump testing
* Strength testing
* Neurocognitive testing Subjects who sustain an injury will undergo repeat testing for comparison to baseline measures.

Further, retrospective chart reviews of past medical history and prospective injury tracking will be collected on all subjects.

DETAILED DESCRIPTION:
The study involves a total of one to three visits, depending on whether an athlete sustains an injury. If an enrolled athlete does not sustain an injury during their athletic season, they will only complete visit 1. If they do, they will complete visits 1, 2, and 3. In total, the expected time requirement is less than 1 hour across the season.

This study will be a two year project in which athletes will be tested around the beginning of their respective sport season.

The PI or Co-I will ask the potential study participant questions regarding inclusion/exclusion criteria. If the potential participant meets all inclusion criteria and no exclusion criteria exist, then the informed consent process can begin. The PI or Co-I will review the informed consent document with the participant. If the participant agrees to be a part of the research study, then the informed consent and authorization form (HIPAA) will be signed electronically.

As part of the 1st Aim of the study: 1 visit, approximately 15 minutes

Information to be collected after consent but does not require the subject to be present:

1. Demographic information, past medical history information and pre-participation examination results from University Athletics athlete health tracking system.
2. Injury occurrence and characteristics during the yearlong season will be tracked and recorded by team athletic trainers and inputted into athlete health tracking system; Such data that will be collected includes but is not limited to: type of injury, location of injury, mechanism of injury, severity of injury, and time missed due to injury.

Initial Pre-season visit (approximately 15 minutes)

All subjects will perform:

1. Sway Sport mobile application assessment tests: reaction time, impulse control, and selective attention (see explanation of study procedures for information on tests). All cognitive testing will be stopped if subject requests to stop. Tests will take approximately 5 minutes.
2. Movement tests: jumping, landing and balance tasks (see explanation of study procedures for information on tests). All physical movement and performance tests will be stopped if subject requests to stop or a significant risk of injury is identified. Tests will take approximately 10 minutes.

Initial pre-season testing should take approximately 15 minutes for actual testing with time requirement of no more than 30 minutes if completing testing in a group setting.

For athletes who sustain non-concussive injuries, standard of care rehab assessments will be collected over the course of recovery and at time of return to play by the treating physical therapist or athletic trainer. These standard of care measures utilized will be up to the rehabilitation provider in their practice and will not add time nor commitment from a research perspective for study participants but may be collected as data to describe injury and recovery characteristics.

As part of the 2nd Aim of the study: 2 additional visits, approximately 15 minutes each Subjects who sustain a concussion, will be identified, and diagnosed by a team physician. As part of the standard University Athletics protocol, these subjects will undergo repeat testing of the following, until they meet satisfactory baseline criteria that is decided upon by the treating physician and athletic trainer.

1. C3Logix neurocognitive testing (see explanation of study procedures for information on tests)
2. Subjective symptom reporting scale as designated by team physician

As part of the study protocol, these subjects will be asked to return for the following repeat testing:

2nd Visit - during week following concussive injury (approximately 15 minutes)

Only subjects that sustain a concussion will perform:

1. Sway Sport mobile application assessment tests: reaction time, impulse control, and selective attention. All cognitive testing will be stopped if subject requests to stop. Tests will take approximately 5 minutes.
2. Movement tests: jumping, landing and balance tasks. All physical movement and performance tests will be stopped if subject requests to stop or a significant risk of injury is identified. Tests will take approximately 10 minutes.

3rd Visit - at time of return to play following concussive injury (approximately 15 minutes)

Only subjects that sustain a concussion will perform:

1. Sway Sport mobile application assessment tests: reaction time, impulse control, and selective attention. All cognitive testing will be stopped if subject requests to stop. Tests will take approximately 5 minutes.
2. Movement tests: jumping, landing and balance tasks. All physical movement and performance tests will be stopped if subject requests to stop or a significant risk of injury is identified. Tests will take approximately 10 minutes.

For athletes who sustain a concussive and/or any non-concussive injuries, standard of care rehab assessments will be collected over the course of recovery and at time of return to play by treating physical therapist or athletic trainer. These standard of care measures utilized will be up to the rehabilitation provider in their practice and will not add time nor commitment from a research perspective for study participants but may be collected as data to describe injury and recovery characteristics.

ELIGIBILITY:
Inclusion Criteria:

* If they are a current National Collegiate Athletics Association (NCAA) student-athlete
* If they are between 17 and 30 years of age - with recent extensions in eligibility requirements for NCAA sports, athletes are participating at increasingly higher ages. Similarly, early enrollees are common and can be included in the study prior to turning 18.

Exclusion Criteria:

* If they are not a current National Collegiate Athletics Association (NCAA) student-athlete
* If they are not between 17 and 30 years of age
* If they are currently experiencing an injury that limits them from completing testing procedures

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Incoming and current NCAA division I collegiate athletes at Texas Christian University
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Movement Tests | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Jumping, landing and balance tasks. Clinical analysis of double limb and single limb jumping, landing and balance on portable force plates. All physical movement and performance tests will be stopped if subject requests to stop or a significant risk of injury is identified. Tests will take approximately 10 minutes.
Sway Neurocognitive Reaction Time Testing | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Sway Sport mobile application assessment test: Reaction time (see explanation of study procedures for information on tests). All cognitive testing will be stopped if subject requests to stop. Tests will take approximately 5 minutes.
Sway Neurocognitive Impulse Control Testing | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Sway Sport mobile application assessment test: Impulse control (see explanation of study procedures for information on tests). All cognitive testing will be stopped if subject requests to stop. Tests will take approximately 5 minutes.
Sway Neurocognitive Cued Stroop Testing | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Sway Sport mobile application assessment test: Selective attention (see explanation of study procedures for information on tests). All cognitive testing will be stopped if subject requests to stop. Tests will take approximately 5 minutes.
Concussion Prospective Injury C3 Logix | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Subjects who sustain a concussion, will be identified, and diagnosed by a team physician. As part of the standard University Athletics protocol, these subjects will undergo repeat testing of the following, until they meet satisfactory baseline criteria that is decided upon by the treating physician and athletic trainer.
  1. C3Logix neurocognitive testing (see explanation of study procedures for information on tests)
Concussion Prospective Injury Tracking - Symptom Reporting | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Subjects who sustain a concussion, will be identified, and diagnosed by a team physician. As part of the standard University Athletics protocol, these subjects will undergo repeat testing of the following, until they meet satisfactory baseline criteria that is decided upon by the treating physician and athletic trainer.
  Collected:
  1. Subjective symptom reporting scale as designated by team physician

SECONDARY OUTCOMES:
Medical History Demographics | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Participant Medical History collected includes:
  Demographic information from University Athletics athlete health tracking system.
Medical History Current Injuries | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Participant Medical History collected includes:
  Current injuries and characteristics from University Athletics athlete health tracking system and Pre-participation physical exam conducted by the University.
Past Medical History Injuries | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Participant Past Medical History collected includes:
  Past injuries and characteristics from University Athletics athlete health tracking system and Pre-participation physical exam conducted by the University.
Medical History Medications | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Participant Medical History collected includes:
  Current medications and supplements from University Athletics athlete health tracking system and Pre-participation physical exam conducted by the University.
Prospective Injury Tracking - Type of Injury | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Injury occurrence and characteristics during the yearlong season will be tracked and recorded by team athletic trainers and inputted into athlete health tracking system:
  Collected:
  Type of injury
Prospective Injury Tracking - Location of Injury | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Injury occurrence and characteristics during the yearlong season will be tracked and recorded by team athletic trainers and inputted into athlete health tracking system:
  Collected:
  Location of injury
Prospective Injury Tracking - Mechanism of Injury | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Injury occurrence and characteristics during the yearlong season will be tracked and recorded by team athletic trainers and inputted into athlete health tracking system:
  Collected:
  Mechanism of injury
Prospective Injury Tracking - Severity of Injury | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Injury occurrence and characteristics during the yearlong season will be tracked and recorded by team athletic trainers and inputted into athlete health tracking system:
  Collected:
  Severity of injury
Prospective Injury Tracking - Time Missed | Baseline testing will occur within the two weeks prior to the start of a sport's season, follow up testing will occur if injury exposure occurs through the study completion (up to 5 years in college setting)
  Injury occurrence and characteristics during the yearlong season will be tracked and recorded by team athletic trainers and inputted into athlete health tracking system:
  Collected:
  Time missed due to injury

CONTACTS AND LOCATIONS:
Overall Officials: Adam C King, Ph.D., Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swanik CB, Covassin T, Stearne DJ, Schatz P. The relationship between neurocognitive function and noncontact anterior cruciate ligament injuries. Am J Sports Med. 2007 Jun;35(6):943-8. doi: 10.1177/0363546507299532. Epub 2007 Mar 16. PMID 17369562
- [Background] Lytle JB, Parikh KB, Tarakemeh A, Vopat BG, Mulcahey MK. Epidemiology of Foot and Ankle Injuries in NCAA Jumping Athletes in the United States During 2009-2014. Orthop J Sports Med. 2021 Apr 16;9(4):2325967121998052. doi: 10.1177/2325967121998052. eCollection 2021 Apr. PMID 33948444
- [Background] Lemoyne J, Poulin C, Richer N, Bussieres A. Analyzing injuries among university-level athletes: prevalence, patterns and risk factors. J Can Chiropr Assoc. 2017 Aug;61(2):88-95. PMID 28928492
- [Background] Lapointe AP, Nolasco LA, Sosnowski A, Andrews E, Martini DN, Palmieri-Smith RM, Gates DH, Broglio SP. Kinematic differences during a jump cut maneuver between individuals with and without a concussion history. Int J Psychophysiol. 2018 Oct;132(Pt A):93-98. doi: 10.1016/j.ijpsycho.2017.08.003. Epub 2017 Aug 14. PMID 28818697
- [Background] Herman DC, Jones D, Harrison A, Moser M, Tillman S, Farmer K, Pass A, Clugston JR, Hernandez J, Chmielewski TL. Concussion May Increase the Risk of Subsequent Lower Extremity Musculoskeletal Injury in Collegiate Athletes. Sports Med. 2017 May;47(5):1003-1010. doi: 10.1007/s40279-016-0607-9. PMID 27544666
- [Background] Chandran A, Boltz AJ, Morris SN, Robison HJ, Nedimyer AK, Collins CL, Register-Mihalik JK. Epidemiology of Concussions in National Collegiate Athletic Association (NCAA) Sports: 2014/15-2018/19. Am J Sports Med. 2022 Feb;50(2):526-536. doi: 10.1177/03635465211060340. Epub 2021 Dec 13. PMID 34898299
- See also: Countermovement Jump Example — https://valdperformance.com/news/understanding-the-countermovement-jump
- See also: Drop Jump Example — https://support.vald.com/hc/en-au/articles/4999913990425-ForceDecks-Test-Drop-Jump-Protocol
- See also: Sway Neurocognitive Simple Reaction Time Testing — https://www.youtube.com/watch?v=RuTK4EbY8p0
- See also: Sway Neurocognitive Impulse Control Testing — https://www.youtube.com/watch?v=NDH7CRP9pYY
- See also: Sway Neurocognitive Selective Attention/Cued Stroop Testing — https://www.linkedin.com/posts/swaymedical_swaytests-cuedstroop-activity-6971499487592681473-j5dR?trk=public_profile_like_view
- See also: C3 Logix Testing — https://www.youtube.com/watch?v=eBcI7Br1c5w